CLINICAL TRIAL: NCT02380508
Title: Evaluation of the Heterologous Effects of Bacille Calmette-Guérin (BCG) Vaccination in Healthy UK Adults
Brief Title: Heterologous Effects of BCG in Healthy UK Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TB038
Record Dates: First submitted 2015-02-03; First posted 2015-03-05 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Tuberculosis
Keywords: BCG study
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): 32 BCG-naïve subjects receiving BCG SSI or BCG Sii at standard dose (2-8x10^5 cfu) via Intradermal route.
  Interventions: Drug: BCG SSI; Drug: BCG Sii
- Group 2 (Experimental): 8-16 control volunteers receiving no vaccination.
  Interventions: Other: No vaccination

INTERVENTIONS:
Drug: BCG SSI — Intradermal injection
  Other Names: Bacille Calmette-Guérin Statens Serum Institute (BCG SSI)
  Arms: Group 1
Other: No vaccination
  Arms: Group 2
Drug: BCG Sii — intradermal injection
  Other Names: Bacille Calmette-Guérin Serum Institute of India
  Arms: Group 1

SUMMARY:
TB038 is a clinical study to assess the non-specific effects of BCG vaccination and gain a better understanding of how the body's immune system reacts to BCG and in turn potentially prevents infection from other bacteria.

DETAILED DESCRIPTION:
Since 1927, it has been observed that BCG-vaccinated neonates have lower all-cause mortality rates. This heterologous or non-specific effect within the first 6-12 months of life has been demonstrated in randomised and observational studies in low income countries with high childhood mortality rates. The most consistent effect is reduced neonatal mortality due to fewer cases of neonatal sepsis, respiratory infection and fever. The main limitation of these studies is the risk of confounding inherent in their cross sectional and observational designs. It is essential that we determine the cogency of this effect, as potential BCG replacement vaccines must be non-inferior to BCG in this regard.

There is a plausible rationale that BCG, a replicating mycobacterium, is capable of inducing non-specific innate immunity, which could induce protection against disease and death from non-mycobacterial infections early in life. For example, intravesical BCG is an effective treatment for bladder cancer, an effect presumed to be non-specific and innate. However, our understanding of the immunological mechanisms involved is incomplete. Data is needed from robust experiments to quantify any causal relationship between infant survival and BCG vaccination. Demonstrating an effect of recent BCG vaccination on the growth of common bacterial pathogens involved in neonatal sepsis, using whole blood in an in-vitro human model, would provide evidence to support a randomised controlled trial in infants in TB high burden countries and would impact on public health vaccination scheduling. In addition it would provide us with an in-vitro model by which to assess future BCG replacement vaccines.

Healthy BCG naïve adults in the UK have been selected for this study because of their low baseline level of anti-mycobacterial immunity and therefore reduced ability to suppress BCG growth. Whilst the target population for the heterologous effects of BCG vaccination is infants, the blood volume required in order to optimise the GIA would not be possible to collect from infants. Therefore by undertaking this work in healthy BCG naïve UK adults we can obtain the blood volumes required for this exploratory work in a population of individuals with a similar background mycobacterial exposure to infants in TB high burden, low income countries.

Volunteers in this study will receive BCG vaccination at the standard dose of 2-8x10^5 cfu. BCG SSI containing Mycobacterium bovis strain Danish 1331 is preferred as it is licensed in the UK for vaccination. However BCG SSI can frequently go into short supply globally with impact on UK supply. In the event of this occurring, BCG vaccine supplied by the Sii (Serum institute of India) will be used instead which contains Mycobacterium bovis BCG strain Moscow 361 I and is on the WHO list of prequalified vaccines. The same strain will be used for all volunteers.

ELIGIBILITY:
Inclusion Criteria:

Volunteers must meet all of the following criteria to enter the study:

* Healthy adult aged 18-45 years
* BCG naïve
* Resident in or near Oxford (for CCTVM and John Warin Ward) or Birmingham (for NIHR WTCRF) for the duration of the study period
* No relevant findings in medical history or on physical examination
* Allow the Investigators to discuss the volunteer's medical history with their GP
* Use effective contraception for the duration of the study period (females only)
* Agreement to refrain from blood donation during the duration of the study and for a period of 3 months after their last visit
* Give written informed consent
* Allow the Investigator to register volunteer details with a confidential database to prevent concurrent entry into clinical trials or studies
* Able and willing (in the Investigator's opinion) to comply with all the study requirements

Exclusion Criteria:

Volunteers must meet none of the following criteria to enter the study:

* Laboratory evidence at screening of latent M. tb infection as indicated by a positive IGRA response
* Clinical, radiological, or laboratory evidence of current active TB disease
* Previous vaccination with BCG, or any candidate TB vaccine
* Within the last year had close household contact with an individual with smear positive pulmonary tuberculosis
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* Concurrent use of long term antibiotic therapy
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the BCG vaccine
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the volunteer in the study
* Positive HBsAg, HCV or HIV antibodies
* Female confirmed pregnant or intention to become pregnant during study period, or currently lactating
* Current involvement in another study or trial that involves regular blood tests or an investigational medicinal product
* Use of an investigational medicinal product or non-registered drug, live vaccine, or investigational medical device for four weeks prior to dosing with the study vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned challenge date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk, or may influence the result of the study, or may affect the volunteer's ability to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Growth inhibition assays | Up to Day 84
  Determine the heterologous effects of BCG vaccination in healthy UK adults using in-vitro Growth Inhibition Assays as a surrogate marker to assess the individuals' capacity to control growth of S. aureus, K. pneumonia, Group B streptococci and E.coli.

SECONDARY OUTCOMES:
Immune response markers | Up to Day 84
  Evaluation of laboratory markers of the immune response that correlate with levels of bacterial growth inhibition identified using the in-vitro GIAs.

OTHER OUTCOMES:
Background levels of S. aureus, K. pneumonia, Group B streptococci and E.coli carriage. | Up to Day 14
  Use of bacterial antibody titres, nasal swab culture and faecal culture to determine background levels of S. aureus, K. pneumonia, Group B streptococci and E.coli carriage in subjects in this study.
Confounding effects of BCG on bacterial growth. | Up tp Day 14
  Use of bacterial antibody titres, nasal swab culture and faecal culture to evaluate confounding effects of BCG on the growth of S. aureus, K. pneumonia, Group B streptococci and E.coli.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Study Director — University of Oxford
Locations (3):
- United Kingdom (3):
  - Centre for Clinical Vaccinology and Tropical Medicine , University of Oxford, Oxford, Oxfordshire
  - Oxford University Hospitals- John Warin Ward, University of Oxford, Oxford, Oxfordshire
  - NIHR Wellcome Trust Clinical Research Facility, University of Birmingham, Birmingham, West Midlands

REFERENCES:
- [Derived] Wilkie M, Tanner R, Wright D, Lopez Ramon R, Beglov J, Riste M, Marshall JL, Harris SA, Bettencourt PJG, Hamidi A, van Diemen PM, Moss P, Satti I, Wyllie D, McShane H. Functional in-vitro evaluation of the non-specific effects of BCG vaccination in a randomised controlled clinical study. Sci Rep. 2022 May 12;12(1):7808. doi: 10.1038/s41598-022-11748-x. PMID 35552463
- See also: Jenner Institute Clinical Trials — http://www.jenner.ac.uk/volunteer